CLINICAL TRIAL: NCT03460496
Title: Transition to Home (TtH) After Preterm Birth: Pilot Testing an Advanced Practice Nurse (APN)-Led Model of Transitional Care
Brief Title: Transition to Home (TtH) After Preterm Birth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Bern University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-01249
Record Dates: First submitted 2018-01-23; First posted 2018-03-09 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Preterm Birth
Keywords: preterm infants; transition to home; advanced practice nurse; cost-analysis
MeSH Terms: conditions — Premature Birth | interventions — Neonatologists; Music Therapy

STUDY DESIGN:
Intervention Model Description: An advanced practice nurse (APN)-led Intervention which focuses on improving parental mental health and well-being, on infant growth and development and on lowering overall costs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APN-led Intervention (Experimental): Intervention group being provided with the interventions described below.
  * Advanced practice nurses' interventions
  * Neonatologists: neonatal outpatient consultation
  * psychological support
  * lactation consultant
  * physiotherapeutic interventions
  * collaboration with social workers
  * music therapy
  * close collaboration with other health care professionals
  * interprofessional roundtable meetings
  Interventions: Behavioral: neonatologists; Behavioral: psychological support; Behavioral: lactation consultant; Behavioral: physiotherapeutic interventions; Behavioral: social workers; Behavioral: music therapy; Behavioral: other health care professionals; Behavioral: interprofessional roundtable meetings; Behavioral: Advanced practice nurses' interventions
- Control, Standard Care (No Intervention): Control group receiving standard care

INTERVENTIONS:
Behavioral: neonatologists — will continue to be contact persons for the APN, even after hospital discharge, and will be available for 3 fixed outpatient consultations with the APN and families that have difficulty getting to a paediatrician, because they live in a rural area with no paediatrician.
  Arms: APN-led Intervention
Behavioral: psychological support — Psychological support will be standard for all families. In a first consultation, psychologist and family will decide about long-term psychological support. They will have at least 3 follow-up consultations during hospital stay and one before discharge; specific psychological interventions will be provided. The aim of the interventions is to re-establish emotional stability and improve the ability of parents to cope with the situation, to prevent parental and family adaptive disorders and child developmental disorders. Support focus on screening for psychological disorders. Techniques include family-centred, holistic interventions (e.g. activating parental resources and coping, crisis intervention, stabilization techniques etc.). Parents will receive outpatient psychological support.
  Arms: APN-led Intervention
Behavioral: lactation consultant — during hospitalization, the lactation consultant will be involved more frequently than during standard care. Breastfeeding support will take a structured approach and will be performed in close collaboration with both parents. The main aims of structured breastfeeding support are strengthen parent-child bonding. Infants will be breastfed according to their needs. Parents will become competent in meeting their child's nutritional needs. After discharge, parents may schedule outpatient breastfeeding consultations.
  Arms: APN-led Intervention
Behavioral: physiotherapeutic interventions — physiotherapeutic interventions will also be structured. The physiotherapist will make an assessment during hospitalization, and decide which physiotherapeutic interventions are necessary. Each family will learn how to handle their premature child in everyday life, based on the child's developmental stage, in a single consultation.
  Arms: APN-led Intervention
Behavioral: social workers — social workers will closely collaborate with the APN within the transitional model. They will be involved with every family and will assist the APN in establishing a network with social and medical services within and outside the clinic. They will also support families in coping with daily life and with their integration into society, family and work. Furthermore, they will give advice on social security issues and on asserting claims as well as clarify financial possibilities.
  Arms: APN-led Intervention
Behavioral: music therapy — music therapy with premature infants and their parents creates a new dimension of contact, and helps stabilize the child and supports their development through music. It also reduces the anxiety of parents, and enhances self-efficacy and makes them more sensitive to their child 74,75, thus enhancing the parent-child relationship. In standard care, music therapy is offered only during hospitalization. In the new model of care, after NICU discharge, the program will offer 10 follow-up sessions at the family's home or in the music therapists' private practice.
  Arms: APN-led Intervention
Behavioral: other health care professionals — the APN will contact and involve other health care professionals, like the family's paediatrician, the outpatient midwife, the community health care nurse or the mother and father counselling as soon as need becomes evident. The APN will help set up meetings between health care professionals and the family, and will keep them up-to-date on the family's situation.
  Arms: APN-led Intervention
Behavioral: interprofessional roundtable meetings — interprofessional roundtable meetings with health care professionals involved in the care of a specific family will be held every two weeks. The meeting is aimed at developing consensus on the best possible support in the care of preterm infants and their families. Parents will be invited to participate in these meetings, led by the APN. The meeting will focus on two family situations, and then determine and initiate supportive interventions in collaboration with the parents.
  Arms: APN-led Intervention
Behavioral: Advanced practice nurses' interventions — The APN will participate in comprehensively planning individual discharge, coordinating services, consulting with other healthcare professionals, assessing needs on a case by case basis, and coaching the family from birth to 6 months after discharge from the NICU. The APN will provide the Newborn Behavioral Observation (NBO), an infant-centred and family-focused method for building relationships, to parents and children, during and after hospitalization. The NBO helps sensitize parents to their infant's competencies and capabilities, teaching them to read their infant's signals and understand their behaviours. It promotes positive interactions between parent and preterm infant. The APN will also offer telephone support and follow-up Visits at home after discharge.
  Arms: APN-led Intervention

SUMMARY:
Preterm birth is associated with significant and often life-long developmental, emotional and financial burdens. Preterm infants face several challenges that continue late into life, including developmental delays, social, and behavioural problems and poor academic performance. Parents also suffer considerable emotional and physical stress which in turn can have a negative impact on the child's development.

In Switzerland, during the transition from hospital to home, there are not many interventions intended to improve mental health outcomes in parents or to promote positive parenting to improve developmental outcomes for the preterm infant. There are also few interventions to reduce associated health care costs.

In order to improve parent and preterm infant outcomes, reduce hospital stay in the neonatal intensive care unit (NICU), lower readmission rates, and avoid unnecessary use of primary care resources a unique, new model of transitional care was developed. The new 'Transition to Home' (TtH) model makes use of well-tested, successful methods of post-discharge care.

The investigators' study will evaluate the organizational and financial feasibility and cost effectiveness of the TtH model for infants born preterm by measuring the impact of an Advanced Practice Nurse (APN)-led intervention at the Children's University Hospital Bern. The intervention focuses on improving parental mental health and well-being, on infant growth and development, and on lowering overall costs. The investigators will gather data and then adapt and test the model within a longitudinal interventional comparative effectiveness study, and prepare it for other Cantons in Switzerland to implement.

DETAILED DESCRIPTION:
In The investigators' model, the APN will participate in comprehensively planning individual discharge, coordinating services, consulting with other healthcare professionals, assessing needs on a case by case basis, and coaching the family from birth to 6 months after discharge from the NICU. The APN will be supported by specialized neonatology nurses; together, they will form the Advanced Nursing Practice Team (ANP Team). Currently, 4 APNs are in training for the project.

The most important tasks of the APN are listed below:

* at birth and during initial hospitalization: first contact of the APN with the family, followed by regular visits, consultations, and educational training for and coordination with other services like lactation consultant, psychologist, social support etc. The APN will conduct family interviews at regular intervals, consult with and train parents on predefined topics in a structured manner while closely collaborating with nursing and medical staff. The APN will take a family-centred approach to making joint decisions. The APN will coordinate health care providers, encourage information flow and collaboration between the professionals as well as organize and manage regular interprofessional exchanges.
* discharge from the hospital: the APN will plan the comprehensive discharge together with parents and the interprofessional team.
* at home: the APN will make systematic follow-up after discharge. The APN will also offer telephone support for requests and answer parent's questions. They will also make follow-up home visits to assess the situation, including assessing physical and mental well-being of parents and infants. The APN will evaluate the interventions the family requested, discuss them with the family, and initiate further services if they are necessary.
* end of the 6 month period: towards the end of the period, the APN will determine, with the parents and other professionals, if the family needs further support, and which specialist would be most appropriate to continue the collaboration with the family.

The role of the interprofessional team:

Within the new model of transitional care, some interprofessional interventions were augmented or adapted.These will be available to families in the intervention group:

Outpatient care by the neonatologist for families that have difficulty getting to a paediatrician, because they live in a rural area with no paediatrician; Standardized psychological support to re-establish emotional stability, improve the ability of parents to cope with the situation and to prevent parental and family adaptive disorders and child developmental disorders; More frequent and standardized involvement of lactation consultant; Standardized involvement of physiotherapy and social workers; Outpatient music therapy.

The APN will contact and involve other health care professionals, like the family's paediatrician, the outpatient midwife, the community health care nurse or the mother and father counselling as soon as need becomes evident. The APN will help set up meetings between health care professionals and the family, and will keep them up-to-date on the family's situation..

Interprofessional roundtable meetings with health care professionals involved in the care of a specific family will be held every two weeks. The meeting is aimed at developing consensus on the best possible support in the care of preterm infants and their families. Parents will be invited to participate in these meetings.

ELIGIBILITY:
Inclusion Criteria:

* Families of preterm infants (between 24 0/7 weeks and 34 6/7 weeks of gestation) born and hospitalized in the University Hospital Bern
* Infants will need to be discharged directly from the Neonatology department, and their parents must reside in Canton Bern, and speak German, French or English.
* For multiple births, all infants will be followed.
* Written informed consent by the parents

Exclusion Criteria:

* Preterm infants with congenital heart malformations and other congenital problems evident at birth

Ages: 24 Weeks to 35 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Parent-child interaction | Once 6 month after discharge
  Parent-child interaction is assessed with the CARE-Index. Three-minute video recordings made in the home setting will be coded by a certified blinded independent coder. The coding procedure focuses on seven aspects of adult and infant behavior. Each aspect of behavior is evaluated separately, for adult and infant, then the scores are summed to generate seven scale scores. For the adult, these are sensitivity, control, and unresponsiveness. For infants they are cooperativeness, compulsiveness, difficultness, and passivity.
  The scores on these scales range from 0-14, with zero sensitivity being dangerously insensitive, 7 being normally sensitive, and 14 being outstandingly sensitive. On the adult sensitivity scale, scores of 5-6 suggest the need for parental education, 3-4 suggests the need for parenting intervention, and 0-2 suggests the need for psychotherapy for the parent.
Parent depressive symptoms | From birth until 6 months after discharge (at 5 time points)
  Depressive symptoms will be assessed with the short version of the 'Allgemeine Depressionsskala' (ADS-K), rated on a 4-point Likert-type scale. The sum score is dichotomized for binary analyses.
Parent anxiety | From birth until 6 months after discharge (at 5 time points)
  Parental anxiety will be assessed with State-Trait Anxiety Inventory (STAI), to measure State Anxiety, and Trait Anxiety. Responses are scored on 4-point forced-choice Likert-type scales.
Parent Posttraumatic Stress Disorder | From birth until 6 months after discharge (at 5 time points)
  PTSD-Checklist (PCL-5) is a 20-item self-report measure that assesses the presence and severity of PTSD symptoms over the past month. Items are rated on a 5-point Likert Scale ranging from 0 (not at all) - 4 (extremely). Items are summed to provide a total severity score (range = 0-80). At total score of 33 or higher indicates the presence of a posttraumatic stress disorder.
Parenting stress | From birth until 6 months after discharge (at 5 time points)
  Parenting stress will be measured with the Parenting Stress Index Short Form (PSI-SF), a self-reporting questionnaire that contains 36 items rated on a 5-point Likert Scale (strongly agree to strongly disagree). Overall parenting stress is indicated by the total stress score. Parents report their level of agreement with 36 items that fall into three subscales (12 items each subscale): Parental distress, parent-child dysfunctional interaction and difficult child. The PSI-SF includes a defensive responding scale (seven items from the Parental Distress scale) that indicates the degree to which the parent might be attempting to deny or minimize problems.
  The raw scores will need to be converted into percentile scores. For each sub-scale a score which falls between the 15th and 80th percentile is considered typical. High scores are those at or above the 85th percentile considering high parenting stress.
Parent self-efficacy | From birth until 6 months after discharge (at 5 time points)
  Tool to measure parenting self-efficacy (TOPSE) is an instrument of 48 statements that encompasses eight dimensions of parenting. The german version of the TOPSE, was reduced to 30 items that encompass five dimensions of parenting (emotion and affection, empathy and understanding, pressures, self-acceptance and learning and knowledge). The items are rated on an 11-point Likert scale.
Infant growth status | From birth until 6 months after discharge
  Growth Status including weight in kg, height in cm and head circumference in cm will be continuously assessed from medical records.
Infant behaviour | Once 6 month after discharge
  Infant temperament, behaviour and self-regulation abilities will be measured used the Infant Behavior Questionnaire-Revised (IBQ-R) short-form at the end of the 6-month study period. IBQ-R consists of 91 items that span 14 scales (Activity Level, Approach, Cuddliness, Distress to Limitations, Duration of Orienting, Falling Reactivity, Fear, High Intensity Pleasure, Low Intensity Pleasure, Perceptual Sensitivity, Sadness, Smiling and Laughter, Soothability and Vocal Reactivity).
Quality of life | From birth until 6 months after discharge (at 3 time points)
  Quality of life will be assessed with the Visual Analog Scale (VAS). Parents will mark a spot along a line from 1 indicating worst possible quality of life to 10 indicating best possible quality of life.
Study burden | Once 6 month after discharge
  Will be evaluated at the end of the study period with a Visual Analog Scale (VAS). Parents will mark a spot along a line from 0 indicating no study burden to 10 indicating highest possible study burden. The VAS will be part of the 6-month questionnaire.
Sleep patterns | From birth until 6 months after discharge
  Sleep patterns will be continuously assessed from medical records.
Self-regulation abilities | From birth until 6 months after discharge
  Self-regulation abilities will be continuously assessed from medical records.

SECONDARY OUTCOMES:
Model evaluation | 6 Month
  Duration, content, and type of contact with all involved healthcare professionals will be documented continuously from hospital and APN records. These will include telephone consultations, home visits and office and hospital visits (including visits to the emergency department). Data will be entered into an Excel sheet for each family.
Cost analysis | 6 Month
  Financial data will be collected for costs incurred during hospital stay as well as post hospital discharge. For the duration of hospital stay the investigators will extract data on length of hospital stay, readmission rates, reason and length of re-hospitalization and all the arising costs from the hospital records. For post-discharge costs, data will be extracted from invoices to patients and a simple questionnaire. The investigators will base cost-effectiveness analyses and cost results on different metrics of outcome measures (Depressive Symptoms, Anxiety, Post-traumatic stress disorders, Parent Child Interaction, Perceived Self-efficacy, etc.).
Infant Nutrition Management and feeding behaviour | From birth until 6 months after discharge
  Infant Nutrition Management including description of what kind of Nutrition the child is getting, in which way the child get's the Nutrition (e.g. breastfeeding) and the nutritional challenges parents are confronted with will be continuously assessed from medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Nelle, PD, Principal Investigator — Insel Gruppe AG, University Hospital Bern; Eva Cignacco, PD, Principal Investigator — Bern University of Applied Sciences
Locations (1):
- Universitätsklinik für Kinderheilkunde Neonatologie Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
The investigators are willing to share IPD but there is no plan description yet available. The investigators will discuss how to develop a plan and the implementation in the upcoming future.